CLINICAL TRIAL: NCT02270138
Title: Movement-to-music Video Program in Decreasing Sedentary Time in Mothers and Children: a Randomized Controlled Trial
Brief Title: An Experimental Study on Music and Sedentariness Among Mothers and Children
Acronym: MovingSound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Sibelius Academy (Unknown); Finnish Institute of Occupational Health (Other); University of Jyvaskyla (Other); Academy of Finland (Other)
Responsible Party: Principal Investigator, Riitta Luoto, Research director, UKK Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 05062014
Record Dates: First submitted 2014-10-02; First posted 2014-10-21 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Sedentary Lifestyle
Keywords: physical activity; music; sedentary lifestyle
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Movement-to-music (Experimental): Three movement-to-music video programs will be used by the participants. First and second videos last about 10 minutes including two songs and their movement preparation. The use of movement-to-music video program will be instructed 10-30 minutes every other day.
  Interventions: Behavioral: Movement-to-music video program
- No movement-to-music (No Intervention): Another group will not receive movement-to-music video during intervention. However, their physical activity will be objectively measured as well.

INTERVENTIONS:
Behavioral: Movement-to-music video program — Three separate movement-to-music video programs will be utilized. Genres of the songs are Children's rock, latin and folk. Range of the tempo is 64-124 beats per minute. The use of movement-to-music video program will be instructed 10-30 minutes every other day.
  Arms: Movement-to-music

SUMMARY:
The aims of the study: Main objective of the current study is to decrease sedentary behavior and increase physical activity among mothers and their offspring by using music-to-movement video program. Primary outcomes of the study are objectively assessed sedentary behavior and physical activity time measured both in minutes and as a proportion of measurement time. Secondary outcomes of the study are quantity and quality of self-reported screen time among mothers and children and motivational quality of music and music-to-movement video. Additional secondary outcomes are mother's weight, workability, mental health and mood. Specific aim is to study effectiveness of intervention with accelerometer use only or with a combination of accelerometer plus music-to-movement video program for mother-child pairs.

Materials and methods: Participants (mother and child -pairs) of the Movement-to-music video program (Moving Sound) -study will be recruited from the cohort of the original Lifestyle, counselling and exercise in maternity care (NELLI) -project from 14 municipalities of Pirkanmaa area. Participants will be randomized in two groups: accelerometer (ACC) vs. accelerometer plus movement-to-music video program (ACC+DVD) groups. Objective measurement of sedentariness and physical activity is based on accelerometer. Information on current health behavior will be based on intervention questionnaires. In the analysis physical activity, sedentary time and body weight of the intervention and control group will be compared. Effects of mother's musical (and PA) background and other mediating factors will be analyzed separately in subgroup analyses.

DETAILED DESCRIPTION:
The aims of the study Quite many people use music during exercise for example while jogging or in the gym. Anyhow some mothers might have difficulties to exercise when they have small children and thereby importance of physical activity at home increases. Consequently, there is a need to perform an experimental study which combines the understanding of the benefits of music, objective physical activity measurement in decreasing sedentariness and thereafter transgenerational obesity.

Main objective of the current study is to decrease sedentary behavior and increase physical activity among mothers and their offspring by using music-to-movement video program.

Specific aim is to study effectiveness of intervention with accelerometer use only or with a combination of accelerometer plus music-to-movement video program for mother-child pairs.

Research questions:

I. Are there changes in sedentary time and physical activity while using accelerometer and movement-to-music video program? Hypothesis: Movement-to-music video program developed for mother-child pairs decrease sedentary time more than wearing accelerometer only. There are no changes in moderate-to-vigorous physical activity, although amount of light intensity physical activity increases.

II. How does motivational effects of music affect to physical activity? Hypothesis: Movement-to-music video motivates mother-child pairs increase physical activity and decrease sedentary behavior.

III. Is there any relationship between mothers' musical background and physical activity/sedentary behavior? Hypothesis: Mothers' musicality motivates them exercise more with video program than mothers' without musical background.

Research methods Accelerometer measures and pretest. Main aim of the project is to reduce sedentariness among women and their children. Accelerometer measures continuously tri-axial acceleration caused by any movement and permits accurate individual assessment of both physical activity and sedentary behavior. Data on physical activity and sedentary behavior will be collected with tri-axial accelerometer (Hookie AM 20, Traxmeet Ltd, Espoo, Finland). The data will be collected in raw mode and analyzed as the mean signal amplitude deviation (MAD) of acceleration, which permits accurate individual assessment of both physical activity and sedentariness. The algorithms used in the present study are based on pilot studies conducted at the UKK Institute.

Accelerometers were pretested with eleven 2-9 years old children. Children did different kind of free movements, play, and games in test track field during one hour. That was done to find out how scurry-like movements appear in accelerometers. Another test in running track tested different speeds from the slow walking to the maximum rate of running. In addition accelerometers piloted with ten 4-7 years children during one week. On the basis of these tests acceleration signal acted as expected.

Movement-to-music DVD production and pretest. There will be three separate movement-to-music video programs prepared by the Sibelius-Academy music education students in the specific course for children's music programs during spring 2014. Directors, Soili Perkiö and Eeva-Leena Pokela are children's music professionals. The student group is called Mutaveijarit (The Mud Mates). Video programs were produced for this study. First and second videos last about 10 minutes including two songs and their movement preparation. There are three songs altogether, because the title song Mutaveijarit is in both tracks. The third video includes all songs together without their movement preparation.

To rate the motivational qualities of these three songs, a panel of 8 physiotherapists (all female) assessed each song by using Brunel Music Rating Inventory-2 (BMRI-2; BMRI-3). Another reason for pretest was to find out the influence of visual stimuli on the responses to the music. BMRI-2 was translated in Finnish by investigators of this study.

Each song was rated by indicating one number between 1 (strongly disagree) and 7 (strongly agree) for six statements about how much the song would motivate a person during exercise. The possible range of scores is 6-42, wherein scores below 24 mean low/oudeterous, middle range 24-35 moderately and scores over 36 mean highly motivating ratings.

Video group (n=4, mean age 41 years, SD 16,2 years) was first watching DVD and assessed all three songs separately using BMRI-2. Then they listened music only (without illustration) and rated the motivational qualities of each song. Music group (n=4, mean age 42,8 years, SD 15,8 years) assessed first only the motivational qualities of the songs. After that music group was watching DVD and appraised the music and illustration together. In addition both groups moved to DVD and rated the motivational qualities of music during movement. All songs were rated moderately motivating (ratings between 31,4 and 34,6).

The rhythm, style, melody, tempo and beat motivated movement more in video group than in music group. Music group assessed sound motivated them more than sound did in video group. During movement rhythm, style, and beat motivated video group more while melody, tempo, and sound motivated music group. As expected in both groups music and picture together motivated movement more than music alone.

Data collection. Objective measurements of sedentary behavior and physical activity of the mothers and their children will be collected at first, second and eighth weeks of the intervention by using accelerometer. Body weight of the mothers will be measured at baseline. Information on current physical activity, screen time, diet, and self-reported weight, as well as information on quality of life will be collected at the baseline by using same questionnaires as in the NELLI 5-years follow-up study (based on one-year follow-up questionnaires of the NELLI cohort). At 2 and 8 weeks after baseline information on physical activity, screen time, self-reported weight and motivation to exercise by using movement-to-music video program will be collected by questionnaires. Information of the children's physical activity and screen time will be collected at baseline, 2nd and 8th weeks after baseline by questionnaires.

Statistical methods. Effect of the intervention will be analyzed following the intention-to-treat principle by comparing the changes in the main outcomes between intervention and control group participants. Multivariate methods corresponding to analysis of covariance and logistic regression will be used. Non-paramet¬ric methods will also be utilized if needed. In the analysis physical activity, sedentary time and body weight of the intervention and control group will be compared. Subgroup analysis in intervention group will be conducted for mother's motivation to exercise with movement-to-music video program and effects of musical background.

Research materials Participants of the Moving Sound -study will be recruited from the cohort of the original NELLI-RTC. Mother and child -pairs (n=837) will be invited to NELLI 5-years follow-up study and to Moving Sound -study from 14 municipalities of Pirkanmaa area. We expect to get involved 30-40 % of the original cohort, which will be 251-335 mother and child -pairs, altogether.

Randomization will be done for 2:2 ratios, which means two mother-child pairs to intervention group per two pairs of control participants. For allocation of the participants an appointment order list for NELLI 5-years follow-up study will be used. Mothers will be randomized to intervention or control group by using sealed envelopes in contact of sampling for NELLI-study.

Power calculations for the study show that approximately 91 mother and child -pairs are needed, if there are 80 % sedentary women at baseline and the anticipated difference in sedentariness is 25 % between the ACC (accelerometer) and ACC + DVD (accelerometer plus movement-to-music video program) groups after intervention. If the anticipated difference between groups is smaller (than 25 %), the number of pairs needed is 135 per group. In this study sedentary women are defined as being sitting or in reclining posture more than 76 % of waking hours.

ELIGIBILITY:
Inclusion Criteria:

* women who have participated to the previous intervention study
* child age between 4 and 7 years

Exclusion Criteria:

* mother and/or child unable to perform physical activity for medical reasons
* mother and/or child unable to use accelerometer as instructed
* no possibility to use DVD player or YouTube-link

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Sedentary lifestyle | Baseline, 8th week
  Objective measurement of sedentary lifestyle with accelerometer; change from baseline in sedentary lifestyle at 8th week

SECONDARY OUTCOMES:
Screen-time | baseline, 8th week
  self-reported quantity and quality of screen time
Motivational quality of music-to-movement video | baseline, 8th week
  Self-reports on questionnaire related to music-to-movement video
Workability | baseline
  Mother's workability, including mental health and mood will be based on self-reported responses to questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Riitta M Luoto, MD, PhD, Principal Investigator — Research director
Locations (1):
- UKK Institute for Health Promotion, Tampere, Finland

REFERENCES:
- [Background] Karageorghis C, Jones L, Stuart DP. Psychological effects of music tempi during exercise. Int J Sports Med. 2008 Jul;29(7):613-9. doi: 10.1055/s-2007-989266. Epub 2007 Nov 30. PMID 18050063
- [Result] Karageorghis CI, Priest DL, Terry PC, Chatzisarantis NL, Lane AM. Redesign and initial validation of an instrument to assess the motivational qualities of music in exercise: the Brunel Music Rating Inventory-2. J Sports Sci. 2006 Aug;24(8):899-909. doi: 10.1080/02640410500298107. PMID 16815785
- [Derived] Tuominen PP, Husu P, Raitanen J, Luoto RM. Rationale and methods for a randomized controlled trial of a movement-to-music video program for decreasing sedentary time among mother-child pairs. BMC Public Health. 2015 Oct 5;15:1016. doi: 10.1186/s12889-015-2347-4. PMID 26438056